CLINICAL TRIAL: NCT03489252
Title: RAMP (Remote Activity Monitoring Pilot): A Feasibility Study Investigating Daily Step and Sleep Data in Combination With Electronic Patient-Reported Outcomes in Adult Patients With Head and Neck Cancer
Brief Title: Remote Activity Monitored by Fitbit Charge 3 in Investigating Daily Step and Sleep Data in Participants With Head and Neck Cancer Undergoing Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17D.653; JT 10656 (Other: JeffTrial Number)
Record Dates: First submitted 2018-03-21; First posted 2018-04-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device Feasibility (Fitbit Charge 3) (Experimental): Participants wear the Fitbit Charge 3 device from the time of CT simulation for RT planning throughout the entire RT course.
  Interventions: Device: Monitoring Device

INTERVENTIONS:
Device: Monitoring Device — Wear Fitbit Charge 3

SUMMARY:
This pilot trial studies remote activity monitored by Fitbit Charge 3 in investigating daily step and sleep data in participants with head and neck cancer who are undergoing radiation therapy. A wearable remote activity tracking device, such as the Fitbit Charge 3, may help to detect early signs of treatment or disease-related symptoms, improve quality of life, decrease emergency room visits, and decrease hospitalizations in participants with head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine compliance with remote activity monitoring (RAM) in patients receiving radiotherapy (RT) or chemoradiotherapy (CRT) for head and neck cancer (HNC).

SECONDARY OBJECTIVES:

I. Evaluate feasibility of recruitment to the Remote Activity Monitoring Pilot (RAMP).

II. Investigate patient acceptability of RAM. III. Evaluate compliance with electronic patient-reported outcomes (ePROs) in this patient population.

IV. Estimate the change in average daily steps associated with a one-unit change in health score as collected on ePRO analysis (analyze associations between RAM data and ePROs).

V. Investigate correlations among step data, quality of life (QOL), and emergency room (ER) visits/hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have head and neck cancer as defined in history and physical
* Patients are eligible to be treated with RT or CRT and plan to start treatment
* Patients are capable of giving informed consent
* Patients must be able to read and/or to speak English
* Patients who are 18 years of age or older
* Women of reproductive potential should have a negative serum or urine pregnancy test within the week prior to radiation CT planning scan

Exclusion Criteria:

* Patients who cannot read or speak English
* Patients who are not candidates for RT/CRT treatment.
* Women of childbearing potential who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Percentage of time patients wear the Fitbit Charge 3 device (compliance) | Through study completion, an average of 3 months
  Daily compliance with remote activity monitoring (RAM) will be defined as wearing the device for 19/24 hours daily (80% daily use). Overall study period compliance will be defined as usage of the device for at least 70% of the days under observation where it should have been worn. The overall study period compliance rate along with a one-sided exact 95% confidence interval will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Voichita Bar-Ad, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States